CLINICAL TRIAL: NCT07148037
Title: Effect of SLC01B1 (rs4149056) Polymorphism on the Efficacy and Tolerability of Atorvastatin in Pakistani Population
Brief Title: Effect of SLC01B1 (rs4149956) Polymorphism on the Efficacy and Tolerability of Atorvastatin in Pakistani Population
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: Riphah/IIMC/IRC/24/1095
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen Description: Venous blood was withdrawn, and DNA extraction was performed using Chelex method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atorvastatin: 10mg once a day for 2 months
  Interventions: Genetic: Atorvastatin

INTERVENTIONS:
Genetic: Atorvastatin — 10mg once a day for 2 months
  Other Names: Statin

SUMMARY:
The goal of this prospective cohort study was to identify the effect of SLC01B1 gene polymorphism in the Pakistani population. The main questions it aims to answer are: To identify polymorphism in SLOC1B1 (rs4149056) in the Pakistani population. To determine the association between SLOC1B1 (rs4149056) polymorphism and the clinical efficacy of atorvastatin To determine the association between SLOC1B1 (rs4149056) polymorphism and the tolerability of atorvastatin

DETAILED DESCRIPTION:
The goal of this prospective cohort study was to identify the effect of SLC01B1 gene polymorphism in the Pakistani population, due to the high prevalence of this variant in the Pakistani Population The main questions it aims to answer are: To identify polymorphism in SLOC1B1 (rs4149056) in the Pakistani population. To determine the association between SLOC1B1 (rs4149056) polymorphism and the clinical efficacy of atorvastatin To determine the association between SLOC1B1 (rs4149056) polymorphism and tolerability of atorvastatin. The participants' blood samples were taken and further genotyping was performed using conventional tetra ARMS PCR. The results were visualized by gel electrophoresis.

ELIGIBILITY:
Inclusion Criteria:

1. Pakistani individuals aged between 40 to 70 years
2. Patients with deranged lipid profile
3. Newly diagnosed patients of dyslipidemia taking atorvastatin (Lipiget) 10mg/day
4. Normal hepatic and renal function

Exclusion Criteria:

1. Patient taking other lipid-lowering medications
2. Moderate and severe systemic diseases
3. Pregnancy
4. Patients taking medications and diet that can interact with atorvastatin
5. Hypothyroidism
6. Recent history of surgical procedure or trauma

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani Population
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
To identify genetic polymorphism in SLOC1B1 in the Pakistani population Genetic polymorphism in SLOC1B1 in the Pakistani population will be assessed by ARMS PCR assay. | 1 month
  To identify genetic polymorphism in SLOC1B1 in the Pakistani population Genetic polymorphism in SLOC1B1 in the Pakistani population will be assessed by ARMS PCR assay.
Lipid profile Lipid profile | 2 months
  Lipid profile Lipid profile will be measured at 0 and on the 56thth day of atorvastatin therapy on a blood sample. LDL cholesterol was categorized as optimal 190mg/dl. Total cholesterol: 240mg/dl = high. HDL cholesterol: 60mg/dl = high. Triglycerides:<150mg/dl were considered optimal, 150-199mg/dl as Borderline high, and 200-500 mg/dl as high
The SAMS-CI tool | 2 months
  The patient will be assessed for tolerability through the myopathy by Statin-associated myopathy (SAM-CI) tool by filling out the questionnaire on days 0, 14,28,42 and 56. The SAMS-CI tool will be used, to record the location, symmetry, and onset of muscle symptoms at day 0, 14,28,42 and 56 of atorvastatin therapy. Patients reporting the presence of muscular pain will be further divided into "Unlikely", "Possible", and "Probable" categories based on their SAMS-CI score.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Waqar, MBBS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hedayatnia M, Asadi Z, Zare-Feyzabadi R, Yaghooti-Khorasani M, Ghazizadeh H, Ghaffarian-Zirak R, Nosrati-Tirkani A, Mohammadi-Bajgiran M, Rohban M, Sadabadi F, Rahimi HR, Ghalandari M, Ghaffari MS, Yousefi A, Pouresmaeili E, Besharatlou MR, Moohebati M, Ferns GA, Esmaily H, Ghayour-Mobarhan M. Dyslipidemia and cardiovascular disease risk among the MASHAD study population. Lipids Health Dis. 2020 Mar 16;19(1):42. doi: 10.1186/s12944-020-01204-y. PMID 32178672
- [Result] Zhang X, Xing L, Jia X, Pang X, Xiang Q, Zhao X, Ma L, Liu Z, Hu K, Wang Z, Cui Y. Comparative Lipid-Lowering/Increasing Efficacy of 7 Statins in Patients with Dyslipidemia, Cardiovascular Diseases, or Diabetes Mellitus: Systematic Review and Network Meta-Analyses of 50 Randomized Controlled Trials. Cardiovasc Ther. 2020 Apr 23;2020:3987065. doi: 10.1155/2020/3987065. eCollection 2020. PMID 32411300
- [Result] Bharath G, Vishnuprabu DP, Preethi L, Nagappan AS, Dhianeshwaran Isravanya RT, Bhaskar LV, Swaminathan N, Munirajan AK. SLCO1B1 and ABCB1 variants synergistically influence the atorvastatin treatment response in South Indian coronary artery disease patients. Pharmacogenomics. 2022 Aug;23(12):683-694. doi: 10.2217/pgs-2022-0044. Epub 2022 Aug 15. PMID 35968761
- [Result] Marin JJG, Serrano MA, Monte MJ, Sanchez-Martin A, Temprano AG, Briz O, Romero MR. Role of Genetic Variations in the Hepatic Handling of Drugs. Int J Mol Sci. 2020 Apr 20;21(8):2884. doi: 10.3390/ijms21082884. PMID 32326111
- [Result] Turongkaravee S, Jittikoon J, Lukkunaprasit T, Sangroongruangsri S, Chaikledkaew U, Thakkinstian A. A systematic review and meta-analysis of genotype-based and individualized data analysis of SLCO1B1 gene and statin-induced myopathy. Pharmacogenomics J. 2021 Jun;21(3):296-307. doi: 10.1038/s41397-021-00208-w. Epub 2021 Feb 19. PMID 33608664